CLINICAL TRIAL: NCT03917459
Title: A Randomized, Double-blind, Active-controlled Study to Assess the Effect of Sacubitril/Valsartan Compared With Enalapril to Improve Erectile Function in Patients With Heart Failure With Reduced Ejection Fraction and Erectile Dysfunction
Brief Title: COmparing arNi and Ace For Improving Erectile Dysfunction in mEN With reduCed Ejection Fraction Heart Failure
Acronym: CONFIDENCE-HF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLCZ696BDE03; 2018-000220-33 (EudraCT Number)
Record Dates: First submitted 2019-04-09; First posted 2019-04-17 (Actual); Results first posted 2024-01-08 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure; Heart Failure, Systolic; Erectile Dysfunction
Keywords: heart failure; systolic heart failure; heart failure with reduced ejection fraction; erectile dysfunction; Enalapril; Enalaprilat; LCZ696; Sacubitril/valsartan
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic; Erectile Dysfunction | interventions — sacubitril and valsartan sodium hydrate drug combination; Enalapril

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LCZ696 (Experimental): LCZ696 200 mg (sacubitril/valsartan 97 mg/103 mg bid)
  Interventions: Drug: LCZ696; Drug: LCZ696 matching placebo
- Enalapril (Active Comparator): Enalapril 10 mg
  Interventions: Drug: Enalapril matching placebo; Drug: Enalapril

INTERVENTIONS:
Drug: LCZ696 — sacubitril/valsartan 200 mg = 97 mg/103 mg bid sacubitril/valsartan film-coated tablets
  Arms: LCZ696
Drug: Enalapril matching placebo — Placebo to Enalapril 10 mg film-coated tablets
  Arms: Enalapril
Drug: Enalapril — Enalapril 10 mg film-coated tablets
  Arms: Enalapril
Drug: LCZ696 matching placebo — Placebo to LCZ696 200 mg = 97 mg/103 mg bid sacubitril/valsartan film-coated tablets
  Arms: LCZ696

SUMMARY:
The purpose of this study was to determine the effect of sacubitril/valsartan (LCZ696) vs. Enalapril on improvement in erectile function and ability in male patients with chronic heart failure with reduced ejection fraction and erectile dysfunction.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the effect of sacubitril/valsartan in improving erectile function in male patients with chronic heart failure (NYHA II) and reduced ejection fraction (HFrEF) and erectile dysfunction (ED). Data from this study was intended to provide a thorough understanding of the impact of sacubitril/valsartan on male sexual function and therefore quality of life.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients with a diagnosis of chronic heart failure (NYHA class II) and reduced ejection fraction (LVEF < 40%)
* Patients must be living in a stable and sexually active heterosexual partnership for at least 6 months prior study start
* Patients must have a mild to moderate erectile dysfunction (determined by using the IIEF-5 questionnaire)
* Patients must be on an ACEI or an ARB at a stable dose for at least 4 weeks prior study start
* Patients must be literate in German

Key Exclusion Criteria:

* History of hypersensitivity to any of the study drugs or its excipients or to drugs of similar chemical classes, ACEIs, ARBs or NEP inhibitors, as well as known or suspected contraindications to the study drugs
* Previous history of intolerance to recommended target doses of ACEIs or ARBs
* Known history of angioedema
* Current acute decompensated HF (exacerbation of chronic HF manifested by signs and symptoms that may require intravenous therapy)
* Symptomatic hypotension
* Impaired renal function
* Penile anatomical defects and Peyronie's disease
* Diabetes mellitus Type I or insulin-dependent Type II
* Known prostate cancer

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- Germany (12):
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Böhlen
  - Novartis Investigative Site, Buchholz in der Nordheide
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Jerichow
  - Novartis Investigative Site, Markkleeberg
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Wermsdorf

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: Plain Language Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1105

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 13 patients were randomized to the LCZ696 group and 14 patients were randomized to the enalapril group. Of these, 12 patients in the LCZ696 group and 13 patients in the enalapril group completed the study. One patient from the LCZ696 group discontinued due to Adverse Event and 1 patient from the enalapril group discontinued due to subject decision.
Pre-assignment Details: A total of 13 patients were randomized to the LCZ696 group and 14 patients were randomized to the enalapril group. Of these, 12 patients in the LCZ696 group and 13 patients in the enalapril group completed the study. One patient from the LCZ696 group discontinued due to Adverse Event and 1 patient from the enalapril group discontinued due to subject decision.
Groups:
- LCZ696: LCZ696 200 mg (sacubitril/valsartan 97 mg/103 mg) bid
- Enalapril: Enalapril 10 mg bid
Period: Overall Study
Arm/Group | LCZ696 | Enalapril
Started | 13 | 14
Completed | 12 | 13
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: A total of 27 patients were included in the Full Analysis Set (FAS) and safety set.
Groups:
- Total: Total of all reporting groups
Arm/Group | LCZ696 | Enalapril | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.5 (9.18) | 66.5 (7.80) | 65.0 (8.47)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender
  Participants
    Female | 0 | 0 | 0
    Male | 13 | 14 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 13 | 14 | 27
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Erectile Function Score Using Index of Erectile Function (IIEF-15)
Description: The International Index of Erectile Function (IIEF-15) was used to assess erectile function in male patients with chronic heart failure. The IIEF-15 is a patient self-reported assessment of erectile dysfunction (ED) and consists of 15 questions assessing different aspects associated with ED. The domain evaluating erectile function consists of items 1, 2, 3, 4, 5 & 15 and its total score was used here. Total score range =1-30. Items 1-5 is 6-point Likert-type scale from '0' (= No sexual activity), '1' (=Almost never or never) to '5' (= Almost always or always). Items 15 is 5-point Likert-type scale from '1' (= very low) to '5 '(= very high). Higher score indicates better outcome
Time Frame: Week 12 (3 months)
Population: All participants who received at least one dose of study treatment and had a valid assessment of the outcome measure
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | LCZ696 | Enalapril
Number analyzed (Participants) | 12 | 13
Scores on a scale | 15.1 (2.15) | 12.2 (2.00)
Statistical Analysis 1: Comparison: LCZ696 vs Enalapril; Test type: Other; p = 0.3432, Mixed Model Repeated Measures (MMRM); LS mean of treatment difference = 2.9, 95% CI 2-sided [-3.29 to 9.01], Standard Error of Mean 2.94

2. Secondary Outcome: Summary of Change From Baseline in Self-reported Frequency of Sexual Activity Per Week
Description: Assessment of early-onset effect and end of study effect, regarding improvement in sexual activity, using patient's self-reported frequency of sexual activity per week. Patient was asked to complete a diary assessing sexual activity on a weekly basis
Time Frame: Baseline, Week 4, Week 12
Population: Full Analysis Set, including all participants who received at least one dose of study treatment
Measure: Mean (Standard Deviation); unit: Activities per week.
Arm/Group | LCZ696 | Enalapril
Number analyzed (Participants) | 13 | 14
Activities per week.
  Week 4:: number analyzed (Participants) | 9 | 11
  Week 4: | -1.6 (1.59) | -1.1 (1.97)
  Week 12:: number analyzed (Participants) | 9 | 8
  Week 12: | -1.4 (3.13) | -2.0 (3.07)

3. Secondary Outcome: Summary of Change From Baseline in NT-proBNP Levels
Description: Change in n-terminal prohormone of brain natriuretic peptide (NT-proBNP) levels compared to baseline assessed at Week 4 and Week 12
Time Frame: Baseline, Week 4, Week 12
Population: Full Analysis Set, including all participants who received at least one dose of study treatment
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | LCZ696 | Enalapril
Number analyzed (Participants) | 13 | 14
pg/mL
  Week 4: number analyzed (Participants) | 13 | 12
  Week 4 | -369.00 [-521.00 to -68.00] | -43.50 [-123.50 to 363.00]
  Week 12: number analyzed (Participants) | 12 | 13
  Week 12 | -208.50 [-1469.00 to 416.50] | -189.00 [-394.00 to 10.00]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of approximately 2 years, 1 month
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment.
Arm/Group | LCZ696 | Enalapril
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/13 | 1/14
Other Adverse Events (participants affected / at risk) | 7/13 | 5/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (N=13) | Enalapril (N=14)
Cardiac arrest (Cardiac disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (N=13) | Enalapril (N=14)
Dental caries (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT03917459/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/59/NCT03917459/SAP_001.pdf